CLINICAL TRIAL: NCT06149936
Title: Efficacy of Excimer Light(308) Therapy for Resistant Alopecia Areata
Brief Title: Excimer Light(308) Therapy for Resistant Alopecia Areata
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hagar Maher, doctor, Assiut University
Other Study IDs: alopecia areata with excimer
Record Dates: First submitted 2021-10-08; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Alopecia Areata
Keywords: excimer light
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: excimer light — Excimer laser using high-dose monochromatic UV radiation

SUMMARY:
This study aimed to evaluate the efficacy and safety of the 308-nm excimer lamp in resistant AA treated with topical minoxidil .

DETAILED DESCRIPTION:
Alopecia areata (AA) is a chronic, nonscarring, T-cell mediated autoimmune disease, presenting with localized or diffuse hair fall in hair-bearing areas. Approximately 1.7% of the population experience an episode of AA during their lifetime. Both sexes are equally affected, and most new cases are recorded below the age of 30 years . Excimer laser using high-dose monochromatic UV radiation can trigger apoptosis and induce immunological suppression through altering cytokine production such as IL-4, IL-10, prostaglandin E2, platelet-activating factor, and cis-urocanic acid. Benefits have only been seen with localized patches of AA, and regrowth of hair occurs only in treated areas .

ELIGIBILITY:
Inclusion Criteria:

* ● Having multiple patches of AA.

  * Duration of alopecia >1 year
  * No topical or systemic treatment for the last 4 months
  * Agreement to regular visits for treatment and follow-up.

Exclusion Criteria:

* ● A single form of AA.

  * Alopecia for <1 year.
  * Being on other modalities of treatment.
  * Treatment within the last 4 months.
  * Photosensitive disorders.
  * Pregnancy or breastfeeding.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: patients take 24 sessions with excimer light for 3 months
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
alopecia areata with ecimer light | 3 months
  evulate patients monthly during treatment with excimer light and minoxidil gel for three months With 20 patients who should completely recovered from alopecia areata.